CLINICAL TRIAL: NCT07116720
Title: The Effect of Unloading Maneuvers During Spinal Flexion Exposure
Brief Title: Unloading Maneuvers During Spinal Flexion Exposure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Primorska (Other)
Responsible Party: Principal Investigator, Matej Voglar, Associate Professor, University of Primorska
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SWE_Flexion3_Intervention
Record Dates: First submitted 2025-08-06; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Occupational Exposure

STUDY DESIGN:
Intervention Model Description: Cross-sectional study with intervention
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Adult participants completing only the spinal flexion protocol
- Intervention group (Experimental): Adult participants performing unloading maneuvers in between the spinal flexion protocol
  Interventions: Other: Unloading maneuvers

INTERVENTIONS:
Other: Unloading maneuvers — Participants will perform unloading maneuvers four times with 15 min of spinal flexion protocol in between. The intervention will include self traction on a box (5 s) and sustained standing trunk extension (8 s). Both maneuvers will be repeated twice at each timepoint.
  Arms: Intervention group

SUMMARY:
An experimental study, which will aim to investigate the acute effects of unloading maneuvers during an intermittent spinal flexion protocol on changes in trunk mechanical and neuromuscular properties.

DETAILED DESCRIPTION:
Our experimental study will include 30 participants. All participants will complete a 60-min intermittent spinal flexion protocol. During rest periods within the protocol, the participants from the intervention group will perform unloading maneuvers for the lumbar spine. Measurements of trunk mechanical and neuromuscular properties. will be performed prior to and following the 60-min protocol.

ELIGIBILITY:
Inclusion Criteria:

* Occupational workers with a predominantly non static job (e.g. combination of sitting and standing)

Exclusion Criteria:

* History of chronic low back pain
* Episode of acute low back pain
* Hip injury in the past six months
* Previous spine, pelvis or hip surgery
* Hypermobility, diagnosed with the Beighton score
* High intensity resistance training (> 75 % of 1 repetition maximum) more than two times a week
* Sporting or recreational activities, that include repetitive spinal flexion or maintenance of a flexed posture (for example cycling or rowing).

Ages: 30 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2025-08-25 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Change in muscle stiffness | 90 minutes
  Muscle stiffness will be measured using ultrasound-based shear wave elastography during prone lying and forward stooping. Erector spinae and multifidus muscle stiffness will be expressed as the shear modulus value in kilopascals.

SECONDARY OUTCOMES:
Change in range of motion | 90 minutes
  Trunk flexion range of motion will be evaluated using Spinal Mouse in maximal trunk flexion while standing.
Change in seated spinal height | 90 minutes
  Seated spinal height will be measured on a custom-developed stadiometer, with the participants in a seated position.
Change in lumbar lordosis angle | 90 minutes
  The lumbar lordosis angle will be evaluated using Spinal Mouse during upright standing.
Change in trunk extension maximal strength | 90 minutes
  Isometric trunk extension peak torque will be assessed on a trunk dynamometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Health Sciences, University of Primorska, Izola, Primorska, Slovenia

IPD SHARING:
Plan to Share IPD: Yes
Coded individual data will be uploaded on public scientific data repository.
Supporting Information: Study Protocol